CLINICAL TRIAL: NCT05029193
Title: Effectiveness of an Online Mindfulness Program for Stroke Survivors and Their Caregivers
Brief Title: Effectiveness of Mindfulness After a Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Harvard University (Other); Chapman University (Other)
Responsible Party: Principal Investigator, Carolee Winstein, Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UP-20-00568-P2
Record Dates: First submitted 2021-08-19; First posted 2021-08-31 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Caregiver Burnout
Keywords: mindfulness; rehabilitation; caregiver; attention to variability
MeSH Terms: conditions — Stroke; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to a mindfulness intervention or a waitlist control. Participants in the waitlist control group will receive the intervention after a 2-month waiting period.
Who Masked: Outcomes Assessor
Masking Description: All outcome measures are self-reported measures administered via online surveys, except for one. The person performing the data analysis will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Stroke survivors - Mindfulness intervention (Experimental): Participants who have had a stroke who are receiving the mindfulness intervention immediately after enrollment (no wait period).
  Interventions: Behavioral: Langerian mindfulness
- Stroke survivors - Waitlist control (No Intervention): Participants who have had a stroke who are assigned to the waitlist.
- Caregivers - Mindfulness intervention (Experimental): Participants caring for someone who have had a stroke and receiving the mindfulness intervention immediately after enrollment (no wait period).
  Interventions: Behavioral: Langerian mindfulness
- Caregivers - Waitlist control (No Intervention): Participants caring for someone who have had a stroke assigned to the waitlist.

INTERVENTIONS:
Behavioral: Langerian mindfulness — A 3-week Langerian mindfulness intervention will be offered entirely online. The purpose of the intervention is: 1) to increase participants' mindfulness, and 2) to encourage participants to change their beliefs about the disability associated with stroke to improve their psychological state. Mindfulness refers to the act of being aware: aware of thoughts, aware of emotions, aware of physical sensations, aware of others. The intervention consists of educational texts, daily exercises, audio recordings and videos. Five different topics related to mindfulness will be introduced throughout the intervention.
  Arms: Caregivers - Mindfulness intervention; Stroke survivors - Mindfulness intervention

SUMMARY:
Mindfulness is promising for individuals with neurological disorders and caregivers to improve psychological well-being. This study aims to determine the extent to which a 3-week online mindfulness intervention will improve quality of life and psychological well-being for chronic stroke survivors and their caregivers, compared to a waitlist control.

DETAILED DESCRIPTION:
Background: The incidence of depression and anxiety is much higher in stroke survivors and their caregivers compared to age-matched peers. Previous work suggests that mindfulness delivered in an online format is promising for both individuals with neurological disorders and caregivers to improve quality of life and psychological well-being.

Aim: This project aims to determine the extent to which a 3-week online mindfulness intervention will improve quality of life and psychological well-being for chronic stroke survivors and their caregivers, compared to a waitlist control. The primary hypothesis is that participants in the mindfulness group will demonstrate greater improvement in quality of life and psychological well-being post-intervention compared to waitlist control participants. The secondary hypothesis is that these improvements will persist for at least 1-month post-intervention.

Methods: This project uses a pragmatic, randomized, waitlist-control trial design with blinded outcome assessment. Participants (stroke survivors and caregivers) are assigned to a 3-week online mindfulness intervention, or a 2-month delayed waitlist. A battery of self-reported outcome measures and clinical tests are administered pre-intervention, post-intervention and at 1-month follow-up. Participants in the waitlist control group are also assessed at enrollment. A sample of 44 stroke survivors and 44 caregivers is targeted. Changes will be measured using a repeated analysis of variance.

Conclusion: The study constitutes the initial step to understand the role of mindfulness exercises delivered remotely and the potential benefit of the intervention for stroke survivors across a wide range of disability level and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivor or caregiver of someone who have had a stroke
* Fluent in English
* Have access to Internet using a computer, a tablet and/or a smart phone.

Exclusion Criteria:

* Severe language impairments
* Participation in regular meditation or a mindfulness program in past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants will not be excluded based on gender.
Enrollment: 29 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the Hospital Anxiety and Depression Scale (HADS) | 2 months
  The HADS assesses depression and anxiety. It is a 14-item scale with 7 items each for anxiety and depression subscales. Each item is scored from 0 to 3, with higher scores indicating higher anxiety or depressive symptoms.
Change from baseline on NIH Toolbox Perceived Stress Survey (PSS) | 2 months
  The PSS assesses perceived stress. It includes 10 items about the occurrence of life stressors scored from 0 (never) to 4 (very often). Higher scores indicate higher perceived stress.
Change from baseline on Single-item Sleep Quality Scale (SQS) | 2 months
  The SQS assesses sleep quality and includes an 11-point visual analogue scale about sleep quality in the past week (0: poor, 10: excellent sleep quality).

SECONDARY OUTCOMES:
Change from baseline on Stroke-specific Quality of Life (SS-QOL) | 2 months
  The SS-QOL assesses health-related quality of life for stroke survivors. It contains 49 items in 12 domains. Items are rated on a 5-point Likert scale from 1 to 5, with higher scores indicating better functioning.
Change from baseline on World Health Organization Quality of Life-BREF (WHOQOL-BREF) | 2 months
  The WHOQOL assesses health-related quality of life and is used in this study to assess caregivers. It comprises 26 questions from 4 domains about health and well-being. The scores are normalized, and higher scores indicate better perceived health and well-being.
Change from baseline on Zarit Burden Interview | 2 months
  The Zarit Burden Interview includes 22 questions about caregiver burden rated from 0 (never) to 4 (nearly always). Higher scores indicate higher perceived burden.
change in the modified Ashworth Scale (elbow) | 2 months
  Measure of spasticity in the flexor and extensor muscles of the elbow. The scores range from 0 to 4, with higher scores indicating more spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Carolee Winstein, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to study protocol, statistical analysis plan and informed consent form on clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The documents will be uploaded by October 2021.